CLINICAL TRIAL: NCT06105632
Title: AN INTERVENTIONAL, OPEN-LABEL, RANDOMIZED, MULTICENTER PHASE 2 STUDY OF PF-07220060 PLUS FULVESTRANT COMPARED TO INVESTIGATOR'S CHOICE OF THERAPY IN PARTICIPANTS AT LEAST 18 YEARS OF AGE WITH HORMONE RECEPTOR-POSITIVE, HER2-NEGATIVE ADVANCED/METASTATIC BREAST CANCER WHOSE DISEASE PROGRESSED AFTER PRIOR CDK 4/6 INHIBITOR-BASED THERAPY (FOURLIGHT-1)
Brief Title: A Study to Learn About the Study Medicine Called PF-07220060 in Combination With Fulvestrant in People With HR-positive, HER2-negative Advanced or Metastatic Breast Cancer Who Progressed After a Prior Line of Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4391022; 2023-506487-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-24; First posted 2023-10-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic Breast Cancer
Keywords: Estrogen receptor positive [ER(+)]; Human epidermal growth factor receptor 2 negative [HER(-)]; ER(+)/HER2(-); Advanced Breast Cancer; Breast tumor; Breast cancer; fulvestrant; everolimus; exemestane; Partial Response+ (PR+); Metastatic breast cancer; Hormone Therapy; Hormone positive breast cancer; Recurrent breast cancer; HR+; HER2-negative; Relapse; Recurrent; Second line treatment.
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — Fulvestrant; Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): PF-07220060 to be taken by mouth as a tablet in combination with fulvestrant (a solution for injection)
  Interventions: Drug: PF-07220060 CDK4 inhibitor; Drug: Fulvestrant
- Arm B (Active Comparator): Investigator's choice of therapy of either:
  * Fulvestrant alone (a solution for injection), or
  * Everolimus in combination with exemestane, both a tablet to be taken by mouth.
  Interventions: Drug: Fulvestrant; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: PF-07220060 CDK4 inhibitor — Experimental
  Arms: Arm A
Drug: Fulvestrant — Experimental and Active comparator
Drug: Everolimus — Active Comparator
  Arms: Arm B
Drug: Exemestane — Active Comparator
  Arms: Arm B

SUMMARY:
The purpose of this study is to learn about the safety and how effective the study medicine (PF-07220060) plus fulvestrant is compared to the study doctor's choice of treatment in people with advanced or metastatic breast cancer. Advanced cancer is the one that is unlikely to be cured or taken care of with treatment. Metastatic cancer is the one that has spread to other parts of the body.

This study is seeking female and male participants who:

* are 18 years of age or older;
* are hormone receptor (HR)-positive and human epidermal growth factor receptor 2 (HER2)-negative;
* have advanced or metastatic breast cancer after taking other treatments before this study;
* have not taken or need to take medications that are not allowed by the study protocol;
* do not have any medical or mental conditions that may increase the risk of study participation.

Half of the participants will take PF-07220060 two times daily by mouth along with fulvestrant. Fulvestrant will be given as a shot into the muscle. The other half will take the study doctor's choice of treatment which can either be:

* Fulvestrant alone taken as shot into the muscle.
* Everolimus along with exemestane taken once daily by mouth.

This study will compare the experiences of participants receiving the study medicine plus fulvestrant to those who are receiving the study doctor's choice of treatment. This will help decide if the study medicine is safe and effective.

Participants will receive study treatment and/or will be in the study until:

* imaging scans (such as an MRI and/or CT) show that their cancer is getting worse.
* the study doctor thinks the participant is no longer benefitting from the study medicine.
* has side effects that become too severe. A side effect is a reaction (expected or unexpected) to a medicine or treatment you take.
* the participant chooses to stop taking part.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast cancer with evidence of locally advanced or metastatic disease, which is not amenable to surgical resection or radiation therapy with curative intent.
* Documented estrogen receptor (ER) and/or progesterone receptor (PR)- positive tumor
* Documented HER2-negative tumor
* Able to provide a sufficient amount of representative formalin fixed, paraffin embedded (FFPE) tumor tissue specimen.
* Must have received CDK4/6i plus NSAI defined per study protocol. There must be documented PD during or after CDK4/6i treatment.
* Measurable disease or non-measurable bone only disease as defined by RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤2.

Exclusion Criteria:

* Any medical or psychiatric condition that may increase the risk of study participation or make the participant inappropriate for the study.
* In visceral crisis at risk of immediately life-threatening complications in the short term.
* Known active uncontrolled or symptomatic central nervous system metastases, carcinomatous meningitis, or leptomeningeal disease.
* Prior treatment with any of the following:
* Everolimus or investigational anti-cancer agents in any setting
* Prior chemotherapy in the advanced setting
* Radiation within 2 weeks of randomization
* Current use or anticipated need for any prohibited food, supplements or concomitant medication(s) (ie, other anti-cancer therapies, other endocrine therapies, growth factors, chronic systemic corticosteroids, strong cytochrome P450 3A4/5 [CYP3A4/5] or uridine 5' diphosphate-glucuronosyltransferase 2B7 [UGT2B7] inhibitors and inducers, direct oral anticoagulants, proton pump inhibitors).
* Inadequate renal function, hepatic dysfunction, or hematologic abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-01-21 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) progression, as determined by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | From Initiation up to 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Time from the date of randomization to the date of death due to any cause up to approximately 3 years
OR by investigator per RECIST v1.1 | Time From randomization date (every 8 weeks during the first 48 weeks and then every 12 weeks) to the date of progression OR death whichever occurs first (up to approximately 2 years)
Duration of Response (DOR) as defined by investigator per RECIST v1.1 | From the date of the first objective response (every 8 weeks during the first 48 weeks and then every 12 week) up to approximately 2 years.
Number of Participants With Clinical Benefit Response (CBR) by investigator per RECIST v1.1 | From randomization date (every 8 weeks during the first 48 weeks and then every 12 weeks) up to approximately 2 years
Number or Patients with Adverse Events (AEs) by Type | From screening until 28 days after the last dose, to approximately 3 years
Number or Patients with AEs by Incidence | From screening until 28 days after the last dose, to approximately 3 years
Number or Patients with AEs by Seriousness | From screening until 28 days after the last dose, to approximately 3 years
Number or Patients with AEs by relationship to study interventions | From screening until 28 days after the last dose, to approximately 3 years
Number of Participants With Abnormal Electrocardiogram (ECG) | From baseline to approximately 2 years
Number of Participants With Laboratory Test Abnormalities | From screening until 28 days after the last dose to approximately 2 years
EQ-5D-5L | Screening Days 1, 15 of Cycle 1 and 2, Day 1 of Cycles 3-6, then Day 1 of every other subsequent Cycle starting with Cycle 8 (eg, Cycles 8, 10, 12, etc) and EoT. Each Cycle is 28 days.
EORTC QLQ | Screening Days 1, 15 of Cycle 1 and 2, Day 1 of Cycles 3-6, then Day 1 of every other subsequent Cycle starting with Cycle 8 (eg, Cycles 8, 10, 12, etc) and EoT. Each Cycle is 28 days.
EORTC QLQ Breast Cancer Module 23 (BR23) | Screening Days 1, 15 of Cycle 1 and 2, Day 1 of Cycles 3-6, then Day 1 of every other subsequent Cycle starting with Cycle 8 (eg, Cycles 8, 10, 12, etc) and EoT. Each Cycle is 28 days.
Ctrough of PF-07220060 | Cycle 1 (Day 15), Cycle 2 (Day 1), and Cycle 3 (Day 1). Each Cycle is 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (153):
- United States (43):
  - UCSF - John Muir Health Cancer Center Berkeley, Berkeley, California
  - Washington Hospital Healthcare System, Fremont, California
  - Hoag Health Center Irvine, Irvine, California
  - Hoag Hospital Irvine, Irvine, California
  - Eisenhower George and Julia Argyros Health Center, La Quinta, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Eisenhower Health Center at South Palm Canyon, Palm Springs, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - UCSF Cancer Center San Mateo, San Mateo, California
  - Saint Vincent's Medical Center (SVMC), Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital (HH), Hartford, Connecticut
  - MidState Medical Center (MMC), Meriden, Connecticut
  - Hartford Healthcare, New Britain, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Hartford HealthCare Cancer Institute at The Hospital of Central Connecticut, Medical Arts Center, Plainville, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - NorthShore University HealthSystem, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - NorthShore University HealthSystem, Highland Park, Illinois
  - Intermountain Health St. Vincent Regional Hospital, Billings, Montana
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana, Billings, Montana
  - Cancer Care Specialists, Reno, Nevada
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Memorial Hermann Cancer Center, Houston, Texas
  - Baylor Scott & White Medical Center - Round Rock, Round Rock, Texas
  - Aurora Health Center - Southern Lakes, Burlington, Wisconsin
  - Aurora Medical Centers - Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Health Center - Kenosha, Kenosha, Wisconsin
  - Aurora Health Center Milwaukee - Good Hope, Milwaukee, Wisconsin
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Medical Center - Summit, Summit, Wisconsin
  - Aurora Cancer Care, Wauwatosa, Wisconsin
- Argentina (11):
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - Organizacion Medica de Investigacion, CABA, Buenos Aires F.D.
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Buenos Aires F.D.
  - Clinica Viedma S. A, Viedma, Río Negro Province
  - Instituto de Oncología de Rosario, Rosario, Santa Fe Province
  - Centro Para la Atención Integral del Paciente Oncologico (CAIPO), San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
  - COE (Centro Oncológico de Excelencia), San Juan
  - Sanatorio Norte, Santiago del Estero
- Australia (2):
  - Macquarie University, North Ryde, New South Wales
  - Icon Cancer Centre Townsville, Rosslea, Queensland
- Brazil (7):
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Pernambuco, Recife, Pernambuco
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Centro de Oncologia - CEON+ - Unidade São Caetano do Sul, São Caetano do Sul, São Paulo
  - Hospital Esperança Recife: Pronto Atendimento 24h, Pernambuco
- Canada (4):
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Jewish General Hospital, Montreal, Quebec
- China (16):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- India (8):
  - Kiran Hospital - Multi Super Speciality Hospital and Research Center, Surat, Gujarat
  - Spandana Oncology Centre (SOC), Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Kims Kingsway Hospital, Nagpur, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
- Israel (3):
  - Rabin Medical Center, Petah Tikva, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
- Japan (15):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma Prefectural Cancer Center, Otashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
- Mexico (8):
  - Boca Clinical Trials Mexico S.C., Guadajalara, Jalisco
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Mexico City
  - Mexico Centre for Clinical Research S.A de C.V, Mexico City, Mexico City
  - COI Centro Oncologico Internacional S.A.P.I. de C.V., Mexico City, Mexico City
  - Filios Alta Medicina S.A. de C.V., Monterrey, Nuevo León
  - Unidad de Investigación en Salud de Chihuahua, S.C., Chihuahua City
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
- South Korea (11):
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-kwangyǒkshi
- Taiwan (7):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (14):
  - Medipol Mega Universite Hastanesi, Stanbul, İ̇stanbul
  - Acibadem Altunizade Hospital, Üsküdar / Stanbul, İ̇stanbul
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Ultramar Medical Imaging Center, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Dicle Üniversitesi, Diyarbakır
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Kocaeli Üniversitesi, Kocaeli
  - Necmettin Erbakan Meram Medical Fac., Konya
  - Samsun Medical Park Hastanesi, Samsun
- United Kingdom (4):
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London, Hammersmith and Fulham
  - Sarah Cannon Research Institute UK, London, London, CITY of
  - The Royal Surrey County Hospital, Guildford
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391022